CLINICAL TRIAL: NCT04657211
Title: Triple thErapy in paTients With COPD Under Real lIve Setting (the TETRIS Study)
Brief Title: Triple Therapy in Chronic Obstructive Pulmonary Disease (COPD) Participants
Acronym: TETRIS
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 214468
Record Dates: First submitted 2020-12-01; First posted 2020-12-08 (Actual); Results first posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD; LABA; LAMA; ICS; TETRIS
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with chronic obstructive pulmonary disease (COPD): Participants with COPD, who will be treated with triple therapy (single inhaler triple therapy [SITT] or multiple inhaler triple therapy [MITT]) for at least 2 but not longer than 48 weeks will be enrolled in this study. No study treatment will be administered during conduct of this study.
  Interventions: Other: Prospective observational cohort study

INTERVENTIONS:
Other: Prospective observational cohort study — prospective observational cohort study

SUMMARY:
TETRIS is a multi-center, prospective observational cohort study. It will include participants with COPD who are on an existing combined treatment of long-acting muscarinic antagonist (LAMA), long-acting beta 2 agonists (LABA) and inhaled corticosteroids (ICS).

DETAILED DESCRIPTION:
COPD is a disabling respiratory disease characterized by airflow obstruction and associated symptoms, including breathing difficulties caused by shortness of breath and wheezing, airway hyperactivity, chronic cough, sputum production, exercise intolerance, and poor quality of life. In accordance with the GOLD (Global Initiative for Chronic Obstructive Lung Disease) recommendations, it is important to assess the characteristics and treatment patterns of participants prior to triple therapy initiation, in order to determine adherence to these guidelines and understand how participants progress to triple therapy. Despite a clearly defined guidance from GOLD treatment recommendations for the initiation and maintenance of triple therapy, treatment changes in Germany, including de-escalation, are often seen in treatment reality. This study is intended to gain a better understanding of what influences the treatment decision of German physicians in primary and secondary care under real life conditions, to elicit the reasons for treatment changes and to describe long-term outcomes with participants initiated on triple therapy over a period of two years. This study will also describe the temporal dynamics of treatment pattern and to unravel potentially complex participant's journeys in different German regions and also to identify and follow-up a variety of 'treatable traits' in COPD participants, which when modified may lead to improved health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Participant is at least 18 years of age at the time of signing the informed consent.
* Participant is on a SITT or MITT for treatment of an obstructive respiratory disease for a period of 6 to 18 weeks prior enrolment with a combination of inhaled LAMA, LABA and ICS either on a triple maintenance treatment or an intermediate triple therapy regime (ICS "on/off" or LAMA "on/off").
* Inclusion criteria for Group A- (treatment by settled general practitioners): Participants are treated according to a physicians diagnosis of COPD.
* Inclusion criteria for Group B and C- (treatment by settled pulmonologists or treatment by outpatient lung centers): Participants have a confirmed physician's diagnosis (diagnosis based on spirometry or body plethysmography) of COPD.
* Participants need to give and be capable of giving signed informed consent form (ICF).

Exclusion Criteria:

* Participant has a diagnosis of pure asthma, without clinical features of COPD.
* Participant has a current diagnosis of lung cancer or lung metastasis.
* Participant has a current primary diagnosis of diffuse pan-bronchiolitis, or a primary diagnosis of bronchiectasis or pulmonary fibrosis or cystic fibrosis or other significant respiratory disorders.
* Participant is currently enrolled or has participated in a study within the last 90 days before signing of consent involving investigational study treatment intervention. If, while enrolled in the present study, the participant enrolls in another study involving investigational study treatment intervention, he/she will be withdrawn from the present study.
* Recent (<= months) major cardiac or pulmonary event (for example myocardial infarction, pulmonary embolism).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study plans to recruit participants with moderate to severe COPD who have been on triple therapy for at least 6 and for a maximum of 18 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 1212 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Hanover, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rohde G, Vogelmeier CF, Beeh KM, Kardos P, Paulsson T, Watz H, Westermayer B, Mohan T, Noorduyn SG, Claussen J. TETRIS - Prospective study to observe clinical outcomes of triple therapy in COPD patients: Up to 12 months interim analysis. Respir Med. 2026 Jan;251:108597. doi: 10.1016/j.rmed.2025.108597. Epub 2025 Dec 17. PMID 41418889
- [Derived] Vogelmeier CF, Beeh KM, Kardos P, Paulsson T, Rohde G, Watz H, Compton C, Mohan T, Claussen J. Baseline patient demographics for TETRIS: a prospective, noninterventional study to characterize the use of triple therapy for COPD in Germany. Ther Adv Respir Dis. 2024 Jan-Dec;18:17534666241287621. doi: 10.1177/17534666241287621. PMID 39436955

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a non-interventional study, it did not include treatment interventions. Data was collected at participant's routine visits.
Pre-assignment Details: Total of 1212 participants were enrolled in this study,however 1196 participants were included in full analysis set(FAS)(as 16 participants were enrolled with incomplete documentation).FAS included all participants who signed Informed Consent Form[ICF],met all inclusion criteria and none of the exclusion criteria, and completed visit1. As pre-specified in protocol and SAP, a combined analysis across all cohorts was performed. Cohorts were used for representative sampling, not separate analyses.
Groups:
- Participants With Chronic Obstructive Pulmonary Disease (COPD): Participants with COPD, who have already been treated with triple therapy (single inhaler triple therapy [SITT] or multiple inhaler triple therapy [MITT]) for at least 2 but not longer than 48 weeks were enrolled in this study. No study treatment was administered during conduct of this study.
Period: Overall Study
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Started | 1212
Full Analysis Set Population | 1196
Safety Analysis Set Population | 1196
Completed | 981
Not Completed | 231
Not completed — Withdrawal by Subject | 21
Not completed — Lost to Follow-up | 113
Not completed — Death | 47
Not completed — Transfer to another institution | 21
Not completed — Other | 29

BASELINE CHARACTERISTICS:
Population: Baseline Characteristic data are reported for the Full Analysis Set which consisted of all participants who signed the ICF, met all inclusion criteria and none of the exclusion criteria, and completed visit 1.
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 1196
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.4 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 634
  Male | 562
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 1196

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Continuously Received Triple Therapy for 6 Months
Description: Percentage of participants who continuously received triple therapy (SITT or MITT) for 6 months from visit 1 (Day 1 of Month 1) have been presented. Percentage values are rounded-off.
Time Frame: From Day 1 (Month 1) up to 6 months
Population: Full Analysis Set included all participants who signed the ICF, met all inclusion criteria and none of the exclusion criteria, and completed visit 1.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 1196
Percentage of participants | 92.5

2. Primary Outcome: Percentage of Participants Who Continuously Received Triple Therapy for 12 Months
Description: Percentage of participants who continuously received triple therapy (SITT or MITT) for 12 months from visit 1 (Day 1 of Month 1) have been presented. Percentage values are rounded-off.
Time Frame: From Day 1 (Month 1) up to 12 months
Population: Full Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 1196
Percentage of participants | 84.4

3. Primary Outcome: Percentage of Participants Who Continuously Received Triple Therapy for 24 Months
Description: Percentage of participants who continuously received triple therapy (SITT or MITT) for 24 months from visit 1 (Day 1 of Month 1) have been presented. Percentage values are rounded-off.
Time Frame: From Day 1 (Month 1) up to 24 months
Population: Full Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 1196
Percentage of participants | 38.5

4. Primary Outcome: Time to Stop Triple Therapy
Description: Time to stop triple therapy refers to the time duration from visit 1 at which a triple therapy (SITT or MITT) was safely and appropriately discontinued because its intended goals had been achieved, or no longer attainable, or risks outweighed the benefits. It was evaluated by Kaplan-Maier analysis.
Time Frame: Up to 24 months
Population: Full Analysis Set.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 1196
Days | 719 [651 to NA] — Less than (<) 75 percent (%) of participants experienced the event within the population. Hence, third-quartile could not be derived.

5. Secondary Outcome: Percentage of Participants With Diagnosis of Asthma at the Age of <40 Years
Description: Percentage of participants with diagnosis of asthma at the age of <40 years have been presented. Data was collected at Baseline visit on Day 1 of inclusion date to the study (Study Day 1). Percentage values are rounded-off.
Time Frame: Baseline (Day 1)
Population: Full Analysis Set. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the Overall Number of Participants Analyzed field.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 8
Percentage of participants | 12.5

6. Secondary Outcome: Percentage of Participants With Peripheral Blood Eosinophils (EOS) Count <100 Cells/uL, 100 to <200 Cells/uL, 200 to <300 Cells/uL and >=300 Cells/uL at Baseline
Description: Percentage of participants with peripheral blood EOS count less than (<) 100 cells per (/) micro liter (uL), 100 to <200 cells/uL, 200 to greater than (>) 300 cells/uL and greater than equal to (>=) 300 cells/uL have been presented. Baseline was considered as Day 1 of inclusion date to the study (Study Day 1). Percentage values are rounded-off.
Time Frame: Baseline (Day 1)
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 94
Percentage of participants
  <100 cells/uL | 23.4
  100 to <200 cells/uL | 26.6
  200 to <300 cells/uL | 19.1
  >=300 cells/uL | 30.9

7. Secondary Outcome: Percentage of Participants With a Physician's Diagnosis of COPD by Site Localization
Description: Percentage of participants with a physician's diagnosis of COPD have been categorized according to the site localization i.e. East, North, South, and West Germany. Data was collected at Baseline visit on Day 1 of inclusion date to the study (Study Day 1). Percentage values are rounded-off.
Time Frame: Baseline (Day 1)
Population: Full Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 1196
Percentage of participants
  East Germany | 23.7
  North Germany | 16.1
  South Germany | 16.1
  West Germany | 44.1

8. Secondary Outcome: Percentage of Participants With a Physician's Diagnosis of COPD by Physicians Group
Description: Percentage of participants with a physician's diagnosis of COPD categorized by pneumologists and general practitioners have been presented. Data was collected at Baseline visit on Day 1 of inclusion date to the study (Study Day 1). Percentage values are rounded-off.
Time Frame: Baseline (Day 1)
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 1196
Percentage of participants
  General practitioners | 38.9
  Pneumologists | 61.1

9. Secondary Outcome: Percentage of Participants With COPD Symptom and Risk Classes (GOLD 1 to 4) at Baseline
Description: COPD was classified using the Global Initiative for Chronic Obstructive Lung Disease (GOLD) criteria. Participants were classified based on symptom and risk of exacerbation, where GOLD 1 (mild COPD), GOLD 2 (moderate COPD), GOLD 3 (severe COPD) and GOLD 4 (very severe COPD). Data for percentage of participants with COPD symptom and risk classes (GOLD 1, GOLD 2, GOLD 3, and GOLD 4) have been presented. Baseline was considered as Day 1 of inclusion date to the study (Study Day 1). Percentage values are rounded-off.
Time Frame: Baseline (Day 1)
Population: Full Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 1196
Percentage of participants
  GOLD 1 | 7.4
  GOLD 2 | 38.0
  GOLD 3 | 28.0
  GOLD 4 | 7.3
  Missing | 19.3

10. Secondary Outcome: Percentage of Participants With COPD Symptom and Risk Classes (GOLD A to D) at Baseline
Description: COPD was classified using the GOLD criteria. Participants are classified based on symptoms and risk of exacerbation, where GOLD A=Few symptoms low risk, GOLD B= More symptoms low risk, GOLD C= Few symptoms high risk and GOLD D= More symptoms high risk. Data for percentage of participants with COPD symptom and risk classes (GOLD A, GOLD B, GOLD C, and GOLD D) have been presented. Baseline was considered as Day 1 of inclusion date to the study (Study Day 1). Percentage values are rounded-off.
Time Frame: Baseline (Day 1)
Population: Full Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 1196
Percentage of participants
  GOLD A | 13.6
  GOLD B | 43.9
  GOLD C | 13.4
  GOLD D | 12.6
  Missing | 16.5

11. Secondary Outcome: Percentage of Participants Who Received Concomitant Respiratory Medication at Months 6, 12 and 24
Description: Percentage of participants with non-missing concomitant respiratory medication received during the study are presented. Percentage of participants were categorized by the substance class of concomitant respiratory medication received by them which included oral glucocorticosteroids, leukotriene receptor antagonist, oral betamimetics, immunotherapy, antibiotics for respiratory indications, and other substances with cardiac or respiratory effects. Percentage values are rounded-off.
Time Frame: At Months 6, 12 and 24
Population: Full Analysis Set. Participants may have provided multiple answers for this question, hence may have contributed to more than one category. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the Overall Number of Participants Analyzed field. 'Number Analyzed' signifies participants evaluable for the specified time points.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 535
Percentage of participants
  Month 6: Oral glucocorticosteroids | 2.6
  Month 6: Leukotriene receptor antagonist | 1.1
  Month 6: Oral betamimetics | 23.4
  Month 6: Immunotherapy | 0.2
  Month 6: Antibiotics for respiratory indications | 1.1
  Month 6: Other substances with cardiac or respiratory effects | 71.6
  Month 12: Oral glucocorticosteroids: number analyzed (Participants) | 524
  Month 12: Oral glucocorticosteroids | 3.2
  Month 12: Leukotriene receptor antagonist: number analyzed (Participants) | 524
  Month 12: Leukotriene receptor antagonist | 1.0
  Month 12: Oral betamimetics: number analyzed (Participants) | 524
  Month 12: Oral betamimetics | 24.0
  Month 12: Immunotherapy: number analyzed (Participants) | 524
  Month 12: Immunotherapy | 0.2
  Month 12: Antibiotics for respiratory indications: number analyzed (Participants) | 524
  Month 12: Antibiotics for respiratory indications | 1.9
  Month 12: Other substances with cardiac or respiratory effects: number analyzed (Participants) | 524
  Month 12: Other substances with cardiac or respiratory effects | 69.7
  Month 24: Oral glucocorticosteroids: number analyzed (Participants) | 492
  Month 24: Oral glucocorticosteroids | 2.6
  Month 24: Leukotriene receptor antagonist: number analyzed (Participants) | 492
  Month 24: Leukotriene receptor antagonist | 1.2
  Month 24: Oral betamimetics: number analyzed (Participants) | 492
  Month 24: Oral betamimetics | 25.6
  Month 24: Immunotherapy: number analyzed (Participants) | 492
  Month 24: Immunotherapy | 0.2
  Month 24: Antibiotics for respiratory indications: number analyzed (Participants) | 492
  Month 24: Antibiotics for respiratory indications | 1.8
  Month 24: Other substances with cardiac or respiratory effects: number analyzed (Participants) | 492
  Month 24: Other substances with cardiac or respiratory effects | 68.5

12. Secondary Outcome: Percentage of Participants by Their Duration of Triple Therapy Before Study Start
Description: Data for percentage of participants by their duration of triple therapy before study start have been presented. Data was categorized into following categories according to duration of triple therapy they received prior to study start: <3 months, 3 to <6 months, >=6 months. Percentage values are rounded-off.
Time Frame: Up to 48 weeks before study start (Day 1 of Month 1)
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 116
Percentage of participants
  <3 months | 31.9
  3 to <6 months | 27.6
  >=6 months | 40.5

13. Secondary Outcome: Percentage of Participants by Their Smoking Status at Months 6, 12 and 24
Description: Percentage of participants were categorized by their smoking status as Lifelong non-smoker, Current smoker and Previous smoker. Percentage values are rounded-off.
Time Frame: At Months 6, 12 and 24
Population: Full Analysis Set. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the Overall Number of Participants Analyzed field. 'Number Analyzed' signifies participants evaluable for the specified time points.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 1091
Percentage of participants
  Month 6: Lifelong non-smoker | 8.8
  Month 6: Current smoker | 37.0
  Month 6: Previous smoker | 54.2
  Month 12: Lifelong non-smoker: number analyzed (Participants) | 1018
  Month 12: Lifelong non-smoker | 8.8
  Month 12: Current smoker: number analyzed (Participants) | 1018
  Month 12: Current smoker | 36.8
  Month 12: Previous smoker: number analyzed (Participants) | 1018
  Month 12: Previous smoker | 54.3
  Month 24: Lifelong non-smoker: number analyzed (Participants) | 930
  Month 24: Lifelong non-smoker | 8.9
  Month 24: Current smoker: number analyzed (Participants) | 930
  Month 24: Current smoker | 36.5
  Month 24: Previous smoker: number analyzed (Participants) | 930
  Month 24: Previous smoker | 54.6

14. Secondary Outcome: Percentage of Participants With a Lifelong Non-smoking History at Baseline
Description: Percentage of participants with a lifelong non-smoking history at Baseline have been presented. Baseline was considered as Day 1 of inclusion date to the study (Study Day 1). Percentage values are rounded-off.
Time Frame: At Baseline (Day 1)
Population: Full Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 1196
Percentage of participants | 8.9

15. Secondary Outcome: Percentage of Participants With Forced Expiratory Volume in 1 Second (FEV1)/Forced Vital Capacity (FVC) Ratio (FEV1/FVC) of <0.7 at Study Enrollment and at 6, 12 and 24 Months
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. FVC is a measure of lung function and is defined as total amount of air that can be exhaled after taking a deep breath. FEV1 and FVC was measured using spirometry. FEV1/FVC ratio was calculated as FEV1/FVC ratio=FEV1/FVC*100. Baseline was considered as Day 1 of inclusion date to the study (Study Day 1). Percentage of participants with FEV1/FVC value <0.7 have been presented. Percentage values are rounded-off.
Time Frame: Baseline (Day 1), Months 6, 12, and 24
Population: as for outcome 13
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 1196
Percentage of participants
  Baseline (Day 1) | 50.4
  Month 6: number analyzed (Participants) | 1091
  Month 6 | 41.5
  Month 12: number analyzed (Participants) | 1018
  Month 12 | 42.8
  Month 24: number analyzed (Participants) | 930
  Month 24 | 42.4

16. Secondary Outcome: Percentage of Participants With Any Moderate/Severe Exacerbation in the 24 Months Prior to Baseline or 3 Months Prior to Each Subsequent On-study Visits at Months 6, 12 and 24
Description: Moderate exacerbations are defined as COPD exacerbations that require either systemic corticosteroids and/or antibiotics. Severe exacerbations are defined as those requiring hospitalization (including intubation and admittance to an intensive care unit) or result in death. Baseline was considered as Day 1 of inclusion date to the study (Study Day 1). Percentage of participants with any moderate/severe exacerbation in the 24 months prior to Baseline or 3 months prior to each subsequent on-study visits at Months 6, 12 and 24 have been presented. Percentage values are rounded-off.
Time Frame: Up to 24 months prior to Baseline (Day 1); Up to 3 months prior to Month 6; Up to 3 months prior to Month 12; Up to 3 months prior to Month 24
Population: as for outcome 13
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 1196
Percentage of participants
  Up to 24 months prior to Baseline | 5.1
  Up to 3 months prior to Month 6: number analyzed (Participants) | 1088
  Up to 3 months prior to Month 6 | 5.6
  Up to 3 months prior to Month 12: number analyzed (Participants) | 1016
  Up to 3 months prior to Month 12 | 8.5
  Up to 3 months prior to Month 24: number analyzed (Participants) | 927
  Up to 3 months prior to Month 24 | 6.8

17. Secondary Outcome: Percentage of Participants With a COPD Assessment Test (CAT) Score <=10, 11-19, >=20 at Baseline and at 6, 12 and 24 Months Documentation
Description: The CAT is a validated measure of health status in COPD. The CAT is an 8-item, patient-completed instrument that covers symptoms such as cough, phlegm, chest tightness, breathlessness, and disease impacts including physical activity, confidence, sleep and energy. Participants rate their experience on a 6-point scale, ranging from 0 (no impairment) to 5 (maximum impairment), higher score indicates greater impairment. A CAT sum score was calculated by summing the non-missing scores of the eight items with a scoring range of 0 (no disease impact) to 40 (maximum disease impact). Higher scores indicated greater disease impact. CAT sum score interpreted as <=10: low impact level, 11-19: Medium impact level, >=20: high impact level. Data for percentage of participants with CAT sum score of <=10, 11-19, and >=20 have been presented. Baseline was considered as Day 1 of inclusion date to the study (Study Day 1). Percentage values are rounded-off.
Time Frame: Baseline (Day 1), Months 6, 12, and 24
Population: as for outcome 13
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 935
Percentage of participants
  Baseline (Day 1): <=10 | 10.7
  Baseline (Day 1): 11-19 | 37.8
  Baseline (Day 1): >=20 | 51.6
  Month 6: <=10: number analyzed (Participants) | 647
  Month 6: <=10 | 14.5
  Month 6: 11-19: number analyzed (Participants) | 647
  Month 6: 11-19 | 48.5
  Month 6: >=20: number analyzed (Participants) | 647
  Month 6: >=20 | 36.9
  Month 12: <=10: number analyzed (Participants) | 544
  Month 12: <=10 | 17.8
  Month 12: 11-19: number analyzed (Participants) | 544
  Month 12: 11-19 | 44.9
  Month 12: >=20: number analyzed (Participants) | 544
  Month 12: >=20 | 37.3
  Month 24: <=10: number analyzed (Participants) | 485
  Month 24: <=10 | 20.6
  Month 24: 11-19: number analyzed (Participants) | 485
  Month 24: 11-19 | 40.8
  Month 24: >=20: number analyzed (Participants) | 485
  Month 24: >=20 | 38.6

18. Secondary Outcome: Percentage of Participants With Peripheral Blood EOS Count of <300 and >=300 Cells/uL at 6, 12 and 24 Months
Description: Percentage of participants with peripheral blood EOS count of <300 cells/uL and >=300 cells/uL have been presented. Percentage values are rounded-off.
Time Frame: At Months 6, 12, and 24
Population: as for outcome 13
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 1091
Percentage of participants
  Month 6: <300 cells/uL | 3.8
  Month 6: >=300 cells/uL | 1.2
  Month 6: Missing | 95.0
  Month 12: <300 cells/uL: number analyzed (Participants) | 1018
  Month 12: <300 cells/uL | 3.5
  Month 12: >=300 cells/uL: number analyzed (Participants) | 1018
  Month 12: >=300 cells/uL | 1.9
  Month 12: Missing: number analyzed (Participants) | 1018
  Month 12: Missing | 94.6
  Month 24: <300 cells/uL: number analyzed (Participants) | 930
  Month 24: <300 cells/uL | 2.9
  Month 24: >=300 cells/uL: number analyzed (Participants) | 930
  Month 24: >=300 cells/uL | 1.3
  Month 24: Missing: number analyzed (Participants) | 930
  Month 24: Missing | 95.8

19. Secondary Outcome: Percentage of Participants With Chronic Bronchitis Phenotype
Description: Chronic bronchitis phenotype is one of the 'treatable traits' in COPD participants, which - when modified - might lead to improved health outcomes. Percentage of participants with chronic bronchitis phenotype have been presented. Percentage values are rounded-off.
Time Frame: Up to 24 months
Population: Full Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 1196
Percentage of participants | 75.5

20. Secondary Outcome: Percentage of Participants With at Least One Switch From Triple Therapy to Long-acting Muscarinic Antagonist (LAMA)/Long-acting Beta Agonist (LABA) From Months 6 to 24
Description: Percentage of participants with at least one switch from triple therapy to LAMA/LABA from Months 6 to 24 have been presented. Percentage values are rounded-off.
Time Frame: Months 6 to 24
Population: Full Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 1196
Percentage of participants | 2.2

21. Secondary Outcome: Percentage of Participants With at Least One Switch From Triple Therapy to Inhaled Corticosteroids (ICS)/LABA From Months 6 to 24
Description: Percentage of participants with at least one switch from triple therapy to ICS/LABA from Months 6 to 24 have been presented. Percentage values are rounded-off.
Time Frame: Months 6 to 24
Population: Full Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 1196
Percentage of participants | 1.5

22. Secondary Outcome: Percentage of Participants With Reasons to Start COPD Triple Therapy in Overall and by Physician Group
Description: Percentage of participants with reasons to start COPD triple therapy in overall participants group have been presented. Reasons to start COPD triple therapy were documented in medical records by physicians. These reasons have been presented in separate categories. Also, data has been presented by type of physician (general practitioners [GP] and pneumologists) who documented these reasons. Percentage values are rounded-off.
Time Frame: Up to 24 months
Population: Full Analysis Set. A participant may have >1 reason to start triple therapy, hence total percentage of participants from different categories (reasons) may not yield 100%. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the Overall Number of Participants Analyzed field. 'Number Analyzed' signifies participants evaluable for the specified time points.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 1196
Percentage of participants
  Overall: Symptomatic despite previous dual therapy with ICS/LABA | 23.4
  Overall: Symptomatic despite previous dual therapy with LAMA/LABA | 52.4
  Overall: Deteriorating quality of life and/or lung function despite long-term therapy | 32.4
  Overall: one or more exacerbations | 15.1
  Overall: Acute exacerbation | 6.7
  Overall: Hospitalization because of major exacerbation/other reason | 3.0
  Overall: Exacerbation prophylaxis | 21.2
  Overall: Participants wish to change medication or device | 20.2
  Overall: Other | 2.3
  Overall: Missing | 0.1
  General practitioners: Symptomatic despite previous dual therapy with ICS/LABA: number analyzed (Participants) | 465
  General practitioners: Symptomatic despite previous dual therapy with ICS/LABA | 24.7
  General practitioners: Symptomatic despite previous dual therapy with LAMA/LABA: number analyzed (Participants) | 465
  General practitioners: Symptomatic despite previous dual therapy with LAMA/LABA | 51.6
  General practitioners: Deteriorating quality of life and/or lung function despite long-term therapy: number analyzed (Participants) | 465
  General practitioners: Deteriorating quality of life and/or lung function despite long-term therapy | 26.2
  General practitioners: one or more exacerbations: number analyzed (Participants) | 465
  General practitioners: one or more exacerbations | 11.0
  General practitioners: Acute exacerbation: number analyzed (Participants) | 465
  General practitioners: Acute exacerbation | 5.8
  General practitioners: Hospitalization because of major exacerbation/other reason: number analyzed (Participants) | 465
  General practitioners: Hospitalization because of major exacerbation/other reason | 2.4
  General practitioners: Exacerbation prophylaxis: number analyzed (Participants) | 465
  General practitioners: Exacerbation prophylaxis | 31.0
  General practitioners: Participants wish to change medication or device: number analyzed (Participants) | 465
  General practitioners: Participants wish to change medication or device | 38.1
  General practitioners: Other: number analyzed (Participants) | 465
  General practitioners: Other | 1.9
  General practitioners: Missing: number analyzed (Participants) | 465
  General practitioners: Missing | 0.2
  Pneumologists: Symptomatic despite previous dual therapy with ICS/LABA: number analyzed (Participants) | 731
  Pneumologists: Symptomatic despite previous dual therapy with ICS/LABA | 22.6
  Pneumologists: Symptomatic despite previous dual therapy with LAMA/LABA: number analyzed (Participants) | 731
  Pneumologists: Symptomatic despite previous dual therapy with LAMA/LABA | 52.9
  Pneumologists: Deteriorating quality of life and/or lung function despite long-term therapy: number analyzed (Participants) | 731
  Pneumologists: Deteriorating quality of life and/or lung function despite long-term therapy | 36.4
  Pneumologists: one or more exacerbations: number analyzed (Participants) | 731
  Pneumologists: one or more exacerbations | 17.8
  Pneumologists: Acute exacerbation: number analyzed (Participants) | 731
  Pneumologists: Acute exacerbation | 7.3
  Pneumologists: Hospitalization because of major exacerbation/other reason: number analyzed (Participants) | 731
  Pneumologists: Hospitalization because of major exacerbation/other reason | 3.4
  Pneumologists: Exacerbation prophylaxis: number analyzed (Participants) | 731
  Pneumologists: Exacerbation prophylaxis | 15.0
  Pneumologists: Participants wish to change medication or device: number analyzed (Participants) | 731
  Pneumologists: Participants wish to change medication or device | 8.8
  Pneumologists: Other: number analyzed (Participants) | 731
  Pneumologists: Other | 2.5
  Pneumologists: Missing: number analyzed (Participants) | 731
  Pneumologists: Missing | 0.0

23. Secondary Outcome: Percentage of Participants With Change From Triple to Dual Therapy and Back to Triple Therapy (at Least One Re-escalation) During a 24-month Observation Period After Study Enrollment (Split by SITT and MITT)
Description: Percentage of participants with change from triple to dual therapy and back to triple therapy (re-escalation) during a 24-month observation period after study enrollment have been presented. Data has been presented in categories split by the type of triple therapy (SITT and MITT) initiated by participants prior to change. Percentage values are rounded-off.
Time Frame: Up to 24 months
Population: as for outcome 13
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 13
Percentage of participants
  Re-escalation: MITT to dual therapy to MITT | 7.7
  Re-escalation: SITT to dual therapy to SITT | 92.3

24. Secondary Outcome: Percentage of Participants With Change From Triple to Dual Therapy and Back to Triple Therapy (at Least One Re-escalation) During a 24-month Observation Period After Study Enrollment (Split by LAMA/LABA, ICS/LABA and ICS/LAMA)
Description: Percentage of participants with change from triple to dual therapy and back to triple therapy (at least one re-escalation) during a 24-month observation period after study enrollment have been presented. Data has been presented in categories split by the type of dual therapy (LAMA/LABA, ICS/LABA and ICS/LAMA) received by participant after change from triple therapy. Percentage values are rounded-off.
Time Frame: Up to 24 months
Population: Full Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 1196
Percentage of participants
  Re-escalation: Triple to LABA/LAMA to Triple | 0.8
  Re-escalation: Triple to LABA/ICS to Triple | 0.3
  Re-escalation: Triple to LAMA/ICS to Triple | 0.0
  No re-escalation | 98.9

25. Secondary Outcome: Percentage of Participants With at Least One Change From MITT to SITT or SITT to MITT During a 24-month Observation Period
Description: Percentage of participants with at least one change in their triple therapy from MITT to SITT or SITT to MITT during a 24-month observation period have been presented. Percentage values are rounded-off.
Time Frame: Up to 24 months
Population: Full Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 1196
Percentage of participants
  MITT to SITT | 3.2
  SITT to MITT | 3.9

26. Secondary Outcome: Percentage of Participants With at Least One Change From SITT to SITT or MITT to MITT During a 24-month Observation Period
Description: Percentage of participants with at least one change within their type of triple therapy - from SITT to SITT or MITT to MITT during a 24-month observation period have been presented. Percentage values are rounded-off.
Time Frame: Up to 24 months
Population: Full Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 1196
Percentage of participants
  SITT to SITT | 2.8
  MITT to MITT | 1.3

27. Secondary Outcome: Percentage of Participants With Change From Once Daily to Twice Daily or Twice Daily to Once Daily Medication
Description: Percentage of participants with change from once daily to twice daily or twice daily to once daily medication has been presented. Percentage values are rounded-off.
Time Frame: Up to 24 months
Population: Full Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 1196
Percentage of participants
  Once daily to twice daily | 3.9
  Twice daily to once daily | 3.2

28. Secondary Outcome: Percentage of Participants With a Change Between Different Inhaler Types
Description: Percentage of participants with a change between different inhaler types have been presented. Percentage values are rounded-off.
Time Frame: Up to 24 months
Population: Full Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 1196
Percentage of participants | 7.8

29. Secondary Outcome: Percentage of Participants With Prespecified Reasons to Change a Triple Therapy (Either MITT or SITT) by Type of Physician Group
Description: Percentage of participants with prespecified reasons to change a triple therapy (TT) (either MITT or SITT) by type of physician group have been presented. Reasons to change a triple therapy were documented in medical records by physicians. These reasons are included in separate categories. Also, data has been presented by type of physician (general practitioners [GP] and pneumologists). Percentage values are rounded-off.
Time Frame: Up to 24 months
Population: Full Analysis Set. A participant may have >1 reason, hence total percentage of participants from different categories (reasons) may not yield 100%. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the Overall Number of Participants Analyzed field. 'Number Analyzed' signifies participants evaluable for the specified time points.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 72
Percentage of participants
  GP: Symptomatic despite previous dual therapy with ICS/LABA: number analyzed (Participants) | 39
  GP: Symptomatic despite previous dual therapy with ICS/LABA | 2.6
  GP: Symptomatic despite previous dual therapy with LAMA/LABA: number analyzed (Participants) | 39
  GP: Symptomatic despite previous dual therapy with LAMA/LABA | 0.0
  GP: Deteriorating quality of life (QoL) and/or lung function despite long-term therapy: number analyzed (Participants) | 39
  GP: Deteriorating quality of life (QoL) and/or lung function despite long-term therapy | 2.6
  GP: One or more exacerbations: number analyzed (Participants) | 39
  GP: One or more exacerbations | 5.1
  GP: Acute exacerbation: number analyzed (Participants) | 39
  GP: Acute exacerbation | 2.6
  GP: Hospitalization because of major exacerbation/other reason: number analyzed (Participants) | 39
  GP: Hospitalization because of major exacerbation/other reason | 5.1
  GP: Exacerbation prophylaxis: number analyzed (Participants) | 39
  GP: Exacerbation prophylaxis | 0.0
  GP: Participants wish to change medication or device: number analyzed (Participants) | 39
  GP: Participants wish to change medication or device | 56.4
  GP: Switching from open TT (MITT, various inhalers) to closed TT (SITT, one inhaler): number analyzed (Participants) | 39
  GP: Switching from open TT (MITT, various inhalers) to closed TT (SITT, one inhaler) | 2.6
  GP: Change from twice daily to once daily: number analyzed (Participants) | 39
  GP: Change from twice daily to once daily | 0.0
  GP: Switching to a different type of inhaler: number analyzed (Participants) | 39
  GP: Switching to a different type of inhaler | 0.0
  GP: Insufficient effectiveness of the previous medication: number analyzed (Participants) | 39
  GP: Insufficient effectiveness of the previous medication | 5.1
  GP: Recommendation of guideline (e.g. discontinuation of ICS): number analyzed (Participants) | 39
  GP: Recommendation of guideline (e.g. discontinuation of ICS) | 0.0
  GP: Recommendation from a referring pulmonologist or acute care clinic: number analyzed (Participants) | 39
  GP: Recommendation from a referring pulmonologist or acute care clinic | 0.0
  GP: Adverse Event: number analyzed (Participants) | 39
  GP: Adverse Event | 0.0
  GP: Symptomatic under existing triple therapy: number analyzed (Participants) | 39
  GP: Symptomatic under existing triple therapy | 35.9
  GP: Other: number analyzed (Participants) | 39
  GP: Other | 7.7
  GP: Missing: number analyzed (Participants) | 39
  GP: Missing | 17.9
  Pneumologists: Symptomatic despite previous dual therapy with ICS/LABA: number analyzed (Participants) | 33
  Pneumologists: Symptomatic despite previous dual therapy with ICS/LABA | 0.0
  Pneumologists: Symptomatic despite previous dual therapy with LAMA/LABA: number analyzed (Participants) | 33
  Pneumologists: Symptomatic despite previous dual therapy with LAMA/LABA | 0.0
  Pneumologists: Deteriorating QoL and/or lung function despite long-term therapy: number analyzed (Participants) | 33
  Pneumologists: Deteriorating QoL and/or lung function despite long-term therapy | 12.1
  Pneumologists: One or more exacerbations: number analyzed (Participants) | 33
  Pneumologists: One or more exacerbations | 6.1
  Pneumologists: Acute exacerbation: number analyzed (Participants) | 33
  Pneumologists: Acute exacerbation | 6.1
  Pneumologists: Hospitalization because of major exacerbation/other reason: number analyzed (Participants) | 33
  Pneumologists: Hospitalization because of major exacerbation/other reason | 0.0
  Pneumologists: Exacerbation prophylaxis: number analyzed (Participants) | 33
  Pneumologists: Exacerbation prophylaxis | 3.0
  Pneumologists: Participants wish to change medication or device: number analyzed (Participants) | 33
  Pneumologists: Participants wish to change medication or device | 21.2
  Pneumologists:Switching from open TT(MITT, various inhalers) to closed TT(SITT, 1 inhaler): number analyzed (Participants) | 33
  Pneumologists:Switching from open TT(MITT, various inhalers) to closed TT(SITT, 1 inhaler) | 6.1
  Pneumologists: Change from twice daily to once daily: number analyzed (Participants) | 33
  Pneumologists: Change from twice daily to once daily | 3.0
  Pneumologists: Switching to a different type of inhaler: number analyzed (Participants) | 33
  Pneumologists: Switching to a different type of inhaler | 9.1
  Pneumologists: Insufficient effectiveness of the previous medication: number analyzed (Participants) | 33
  Pneumologists: Insufficient effectiveness of the previous medication | 6.1
  Pneumologists: Recommendation of guideline (e.g. discontinuation of ICS): number analyzed (Participants) | 33
  Pneumologists: Recommendation of guideline (e.g. discontinuation of ICS) | 0.0
  Pneumologists: Recommendation from a referring pulmonologist or acute care clinic: number analyzed (Participants) | 33
  Pneumologists: Recommendation from a referring pulmonologist or acute care clinic | 0.0
  Pneumologists: Adverse Event: number analyzed (Participants) | 33
  Pneumologists: Adverse Event | 3.0
  Pneumologists: Symptomatic under existing triple therapy: number analyzed (Participants) | 33
  Pneumologists: Symptomatic under existing triple therapy | 24.2
  Pneumologists: Other: number analyzed (Participants) | 33
  Pneumologists: Other | 9.1
  Pneumologists: Missing: number analyzed (Participants) | 33
  Pneumologists: Missing | 24.2

30. Secondary Outcome: Percentage of Participants With Reasons for Change in Their Triple Therapy to Another Triple Therapy in Overall Participants
Description: Percentage of participants with reasons for change in their triple therapy to another triple therapy in overall participants group have been presented. Reasons for change in triple therapy to another triple therapy were documented in medical records by physician. These reasons are included in separate categories. Percentage values are rounded-off.
Time Frame: Up to 24 months
Population: Full Analysis Set. A participant may have >1 reason, hence total percentage of participants from different categories (reasons) may not yield 100%. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the Overall Number of Participants Analyzed field.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 72
Percentage of participants
  Symptomatic despite previous dual therapy with ICS/LABA | 1.4
  Symptomatic despite previous dual therapy with LAMA/LABA | 0.0
  Deteriorating quality of life (QoL) and/or lung function despite long-term therapy | 6.9
  One or more exacerbations | 5.6
  Acute exacerbation | 4.2
  Hospitalization because of major exacerbation/other reason | 2.8
  Exacerbation prophylaxis | 1.4
  Participants wish to change medication or device | 40.3
  Switching from open TT (MITT, various inhalers) to closed TT (SITT, one inhaler) | 4.2
  Change from twice daily to once daily | 1.4
  Switching to a different type of inhaler | 4.2
  Insufficient effectiveness of the previous medication | 5.6
  Recommendation of guideline (e.g. discontinuation of ICS) | 0.0
  Recommendation from a referring pulmonologist or acute care clinic | 0.0
  Adverse Event | 1.4
  Symptomatic under existing triple therapy | 30.6
  Other | 8.3
  Missing | 20.8

31. Secondary Outcome: Percentage of Participants With Reasons for Change From Triple Therapy to Therapy De-escalation
Description: Percentage of participants with reasons for change from triple therapy to therapy de-escalation in overall participants group have been presented. A participant was classified as de-escalation, if there was at least one change from triple therapy to a therapy with just two components within the first 365 days of observation. Reasons for change from triple therapy to therapy de-escalation were documented in medical records by physicians. These reasons are included in separate categories. Percentage values are rounded-off.
Time Frame: Up to 24 months
Population: as for outcome 30
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 27
Percentage of participants
  Symptomatic despite previous dual therapy with ICS/LABA | 0.0
  Symptomatic despite previous dual therapy with LAMA/LABA | 0.0
  Deteriorating quality of life (QoL) and/or lung function despite long-term therapy | 7.4
  One or more exacerbations | 3.7
  Acute exacerbation | 0.0
  Hospitalization because of major exacerbation/other reason | 0.0
  Exacerbation prophylaxis | 3.7
  Participants wish to change medication or device | 63.0
  Switching from open TT (MITT, various inhalers) to closed TT (SITT, one inhaler) | 0.0
  Change from twice daily to once daily | 3.7
  Switching to a different type of inhaler | 3.7
  Insufficient effectiveness of the previous medication | 3.7
  Recommendation of guideline (e.g. discontinuation of ICS) | 0.0
  Recommendation from a referring pulmonologist or acute care clinic | 3.7
  Adverse Event | 3.7
  Symptomatic under existing triple therapy | 3.7
  Other | 7.4
  Missing | 22.2

32. Secondary Outcome: Percentage of Participants With Reasons to Change De-escalated Therapy Back to Triple Therapy
Description: Percentage of participants with reasons to change de-escalated therapy back to triple therapy in overall participants group have been presented. A participant was classified as de-escalation, if there was at least one change from triple therapy to a therapy with just two components within the first 365 days of observation. Reasons to change de-escalated therapy back to triple therapy were documented in medical records by physicians. These reasons are included in separate categories. Percentage values are rounded-off.
Time Frame: Up to 24 months
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 10
Percentage of participants
  Symptomatic despite previous dual therapy with ICS/LABA | 0.0
  Symptomatic despite previous dual therapy with LAMA/LABA | 0.0
  Deteriorating quality of life (QoL) and/or lung function despite long-term therapy | 10.0
  One or more exacerbations | 0.0
  Acute exacerbation | 10.0
  Hospitalization because of major exacerbation/other reason | 0.0
  Exacerbation prophylaxis | 0.0
  Participants wish to change medication or device | 20.0
  Switching from open TT (MITT, various inhalers) to closed TT (SITT, one inhaler) | 0.0
  Change from twice daily to once daily | 0.0
  Switching to a different type of inhaler | 0.0
  Insufficient effectiveness of the previous medication | 10.0
  Recommendation of guideline (e.g. discontinuation of ICS) | 0.0
  Recommendation from a referring pulmonologist or acute care clinic | 20.0
  Adverse Event | 0.0
  Symptomatic under existing triple therapy | 0.0
  Other | 10.0
  Missing | 20.0

33. Secondary Outcome: Mean Annual Rate of Moderate and/or Severe Exacerbations in Overall Participants and by Their Peripheral Blood Eosinophil Count, Smoking Status and Asthma History
Description: The annual rate of moderate and severe chronic obstructive pulmonary disease (COPD) exacerbations during the study period (per participant per year) was assessed. Annualized rate of moderate and severe exacerbations was calculated as Annual exacerbation rate = total number of moderate or severe exacerbation/total person years. Moderate exacerbations are defined as COPD exacerbations that require either systemic corticosteroids and/or antibiotics. Severe exacerbations are defined as those requiring hospitalization (including intubation and admittance to an intensive care unit) or result in death. Data for mean annual rate of moderate and/or severe exacerbations is presented for overall participants, and by their peripheral EOS count (missing, <300 and >=300 cells/uL), smoking status (Lifelong non-smoker, Current and previous smoker) and asthma history (missing, yes, no and unknown).
Time Frame: Up to 24 months
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Exacerbations per participant per year
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 1196
Exacerbations per participant per year
  Overall | 0.156 (0.465)
  Smoking status: Lifelong non-smoker: number analyzed (Participants) | 106
  Smoking status: Lifelong non-smoker | 0.128 (0.458)
  Smoking status: Current smoker: number analyzed (Participants) | 454
  Smoking status: Current smoker | 0.102 (0.296)
  Smoking status: Previous smoker: number analyzed (Participants) | 636
  Smoking status: Previous smoker | 0.199 (0.553)
  Eosinophil count: <300 cells/uL: number analyzed (Participants) | 65
  Eosinophil count: <300 cells/uL | 0.445 (0.923)
  Eosinophil count: >=300 cells/uL: number analyzed (Participants) | 29
  Eosinophil count: >=300 cells/uL | 0.238 (0.671)
  Eosinophil count: Missing: number analyzed (Participants) | 1102
  Eosinophil count: Missing | 0.145 (0.433)
  Asthma history: No: number analyzed (Participants) | 923
  Asthma history: No | 0.152 (0.446)
  Asthma history: Yes: number analyzed (Participants) | 193
  Asthma history: Yes | 0.162 (0.439)
  Asthma history: Missing: number analyzed (Participants) | 14
  Asthma history: Missing | 0.176 (0.523)
  Asthma history: Unknown: number analyzed (Participants) | 66
  Asthma history: Unknown | 0.161 (0.568)

34. Secondary Outcome: Mean Annual Rate of Hospitalizations Due to Severe Exacerbations
Description: Severe exacerbations are defined as those requiring hospitalization (including intubation and admittance to an intensive care unit) or result in death. Annualized rate of hospitalization due to severe exacerbations was calculated as Annual hospitalization rate equal to (=) number of hospitalizations due to severe exacerbations divided by (/) total person years.
Time Frame: Up to 24 months
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Hospitalization per participant per year
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 1196
Hospitalization per participant per year | 0.058 (0.303)

35. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) in Overall Participants and by Their Peripheral Blood Eosinophil Count, Smoking Status and Asthma History at Month 6
Description: FEV1 is a measure of lung function and is defined as the volume of air that can be forced out in one second after taking a deep breath. FEV1 was measured electronically by spirometry. Baseline was considered as Day 1 of inclusion date to the study (Study Day 1). Change from Baseline was calculated as the value at Month 6 minus the value at Baseline. Data for change from Baseline in FEV1 is presented for overall participants, and by their peripheral blood eosinophil count (missing, <300 and >=300 cells/uL), smoking history (Lifelong non-smoker, Current and previous smoker) and asthma history (missing, yes, no and unknown).
Time Frame: Baseline (Day 1) and at Month 6
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 717
Liter
  Overall | 0.01 (0.38)
  Peripheral blood EOS: <300 cells/uL: number analyzed (Participants) | 33
  Peripheral blood EOS: <300 cells/uL | -0.04 (0.46)
  Peripheral blood EOS: >=300 cells/uL: number analyzed (Participants) | 20
  Peripheral blood EOS: >=300 cells/uL | 0.00 (0.28)
  Peripheral blood EOS: Missing: number analyzed (Participants) | 664
  Peripheral blood EOS: Missing | 0.02 (0.37)
  Smoking history: Lifelong non-smoker: number analyzed (Participants) | 62
  Smoking history: Lifelong non-smoker | -0.04 (0.39)
  Smoking history: Current smoker: number analyzed (Participants) | 269
  Smoking history: Current smoker | 0.02 (0.39)
  Smoking history: Previous smoker: number analyzed (Participants) | 386
  Smoking history: Previous smoker | 0.02 (0.36)
  Asthma history: No: number analyzed (Participants) | 588
  Asthma history: No | 0.00 (0.37)
  Asthma history: Yes: number analyzed (Participants) | 16
  Asthma history: Yes | 0.08 (0.28)
  Asthma history: Unknown: number analyzed (Participants) | 9
  Asthma history: Unknown | 0.37 (0.53)
  Asthma history: Missing: number analyzed (Participants) | 104
  Asthma history: Missing | 0.05 (0.38)

36. Secondary Outcome: Change From Baseline in FEV1 in Overall Participants and by Their Peripheral Blood Eosinophil Count, Smoking Status and Asthma History at Month 12
Description: FEV1 is a measure of lung function and is defined as the volume of air that can be forced out in one second after taking a deep breath. FEV1 was measured electronically by spirometry. Baseline was considered as Day 1 of inclusion date to the study (Study Day 1). Change from Baseline was calculated as the value at Month 12 minus the value at Baseline. Data for change from Baseline in FEV1 is presented for overall participants, and by their peripheral blood eosinophil count (missing, <300 and >=300 cells/uL), smoking history (Lifelong non-smoker, Current and previous smoker) and asthma history (missing, yes, no and unknown).
Time Frame: Baseline (Day 1) and at Month 12
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 709
Liter
  Overall | 0.02 (0.48)
  Peripheral blood EOS: <300 cells/uL: number analyzed (Participants) | 31
  Peripheral blood EOS: <300 cells/uL | -0.07 (0.52)
  Peripheral blood EOS: >=300 cells/uL: number analyzed (Participants) | 18
  Peripheral blood EOS: >=300 cells/uL | -0.16 (0.36)
  Peripheral blood EOS: Missing: number analyzed (Participants) | 660
  Peripheral blood EOS: Missing | 0.03 (0.48)
  Smoking history: Lifelong non-smoker: number analyzed (Participants) | 61
  Smoking history: Lifelong non-smoker | -0.01 (0.47)
  Smoking history: Current smoker: number analyzed (Participants) | 252
  Smoking history: Current smoker | 0.04 (0.55)
  Smoking history: Previous smoker: number analyzed (Participants) | 396
  Smoking history: Previous smoker | 0.01 (0.44)
  Asthma history: No: number analyzed (Participants) | 569
  Asthma history: No | -0.02 (0.42)
  Asthma history: Yes: number analyzed (Participants) | 16
  Asthma history: Yes | 0.23 (0.81)
  Asthma history: Unknown: number analyzed (Participants) | 21
  Asthma history: Unknown | 0.78 (0.87)
  Asthma history: Missing: number analyzed (Participants) | 103
  Asthma history: Missing | 0.08 (0.48)

37. Secondary Outcome: Change From Baseline in FEV1 in Overall Participants and by Their Peripheral Blood Eosinophil Count, Smoking Status and Asthma History at Month 24
Description: FEV1 is a measure of lung function and is defined as the volume of air that can be forced out in one second after taking a deep breath. FEV1 was measured electronically by spirometry. Baseline was considered as Day 1 of inclusion date to the study (Study Day 1). Change from Baseline was calculated as the value at Month 24 minus the value at Baseline. Data for change from Baseline in FEV1 is presented for overall participants, and by their peripheral blood eosinophil count (missing, <300 and >=300 cells/uL), smoking history (Lifelong non-smoker, Current and previous smoker) and asthma history (missing, yes, no and unknown).
Time Frame: Baseline (Day 1) and at Month 24
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 657
Liter
  Overall | 0.00 (0.52)
  Peripheral blood EOS: <300 cells/uL: number analyzed (Participants) | 32
  Peripheral blood EOS: <300 cells/uL | 0.04 (0.56)
  Peripheral blood EOS: >=300 cells/uL: number analyzed (Participants) | 18
  Peripheral blood EOS: >=300 cells/uL | -0.13 (0.59)
  Peripheral blood EOS: Missing: number analyzed (Participants) | 607
  Peripheral blood EOS: Missing | 0.00 (0.51)
  Smoking history: Lifelong non-smoker: number analyzed (Participants) | 59
  Smoking history: Lifelong non-smoker | -0.04 (0.52)
  Smoking history: Current smoker: number analyzed (Participants) | 246
  Smoking history: Current smoker | 0.03 (0.59)
  Smoking history: Previous smoker: number analyzed (Participants) | 352
  Smoking history: Previous smoker | -0.01 (0.46)
  Asthma history: No: number analyzed (Participants) | 524
  Asthma history: No | -0.04 (0.47)
  Asthma history: Yes: number analyzed (Participants) | 14
  Asthma history: Yes | 0.15 (0.82)
  Asthma history: Unknown: number analyzed (Participants) | 20
  Asthma history: Unknown | 0.85 (0.74)
  Asthma history: Missing: number analyzed (Participants) | 99
  Asthma history: Missing | 0.02 (0.49)

38. Secondary Outcome: Change From Baseline in Forced Vital Capacity (FVC) in Overall Participants and by Their Peripheral Blood Eosinophil Count, Smoking Status and Asthma History at Month 6
Description: FVC is a measure of lung function and is defined as total amount of air that can be exhaled after taking a deep breath. FVC was measured using spirometry. Baseline was considered as Day 1 of inclusion date to the study (Study Day 1). Change from Baseline was calculated as the value at Month 6 minus the value at Baseline. Data for change from Baseline in FVC is presented for overall participants, and by their peripheral blood eosinophil count (missing, <300 and >=300 cells/uL), smoking history (Lifelong non-smoker, Current and previous smoker) and asthma history (missing, yes, no and unknown).
Time Frame: Baseline (Day 1) and at Month 6
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 591
Liter
  Overall | 0.02 (0.46)
  Peripheral blood EOS: <300 cells/uL: number analyzed (Participants) | 28
  Peripheral blood EOS: <300 cells/uL | -0.03 (0.58)
  Peripheral blood EOS: >=300 cells/uL: number analyzed (Participants) | 18
  Peripheral blood EOS: >=300 cells/uL | -0.06 (0.29)
  Peripheral blood EOS: Missing: number analyzed (Participants) | 545
  Peripheral blood EOS: Missing | 0.02 (0.45)
  Smoking history: Lifelong non-smoker: number analyzed (Participants) | 41
  Smoking history: Lifelong non-smoker | 0.02 (0.39)
  Smoking history: Current smoker: number analyzed (Participants) | 214
  Smoking history: Current smoker | 0.01 (0.46)
  Smoking history: Previous smoker: number analyzed (Participants) | 336
  Smoking history: Previous smoker | 0.02 (0.46)
  Asthma history: No: number analyzed (Participants) | 481
  Asthma history: No | 0.02 (0.44)
  Asthma history: Yes: number analyzed (Participants) | 13
  Asthma history: Yes | 0.00 (0.45)
  Asthma history: Unknown: number analyzed (Participants) | 7
  Asthma history: Unknown | 0.17 (0.35)
  Asthma history: Missing: number analyzed (Participants) | 90
  Asthma history: Missing | 0.01 (0.53)

39. Secondary Outcome: Change From Baseline in FVC in Overall Participants and by Their Peripheral Blood Eosinophil Count, Smoking Status and Asthma History at Month 12
Description: FVC is a measure of lung function and is defined as total amount of air that can be exhaled after taking a deep breath. FVC was measured using spirometry. Baseline was considered as Day 1 of inclusion date to the study (Study Day 1). Change from Baseline was calculated as the value at Month 12 minus the value at Baseline. Data for change from Baseline in FVC is presented for overall participants, and by their peripheral blood eosinophil count (missing, <300 and >=300 cells/uL), smoking history (Lifelong non-smoker, Current and previous smoker) and asthma history (missing, yes, no and unknown).
Time Frame: Baseline (Day 1) and at Month 12
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 577
Liter
  Overall | -0.02 (0.53)
  Peripheral blood EOS: <300 cells/uL: number analyzed (Participants) | 24
  Peripheral blood EOS: <300 cells/uL | -0.05 (0.70)
  Peripheral blood EOS: >=300 cells/uL: number analyzed (Participants) | 16
  Peripheral blood EOS: >=300 cells/uL | -0.24 (0.46)
  Peripheral blood EOS: Missing: number analyzed (Participants) | 537
  Peripheral blood EOS: Missing | -0.01 (0.52)
  Smoking history: Lifelong non-smoker: number analyzed (Participants) | 44
  Smoking history: Lifelong non-smoker | 0.22 (0.41)
  Smoking history: Current smoker: number analyzed (Participants) | 192
  Smoking history: Current smoker | -0.05 (0.49)
  Smoking history: Previous smoker: number analyzed (Participants) | 341
  Smoking history: Previous smoker | -0.03 (0.55)
  Asthma history: No: number analyzed (Participants) | 469
  Asthma history: No | -0.03 (0.52)
  Asthma history: Yes: number analyzed (Participants) | 12
  Asthma history: Yes | -0.12 (0.62)
  Asthma history: Unknown: number analyzed (Participants) | 9
  Asthma history: Unknown | 0.07 (0.58)
  Asthma history: Missing: number analyzed (Participants) | 87
  Asthma history: Missing | 0.00 (0.57)

40. Secondary Outcome: Change From Baseline in FVC in Overall Participants and by Their Peripheral Blood Eosinophil Count, Smoking Status and Asthma History at Month 24
Description: FVC is a measure of lung function and is defined as total amount of air that can be exhaled after taking a deep breath. FVC was measured using spirometry. Baseline was considered as Day 1 of inclusion date to the study (Study Day 1). Change from Baseline was calculated as the value at Month 24 minus the value at Baseline. Data for change from Baseline in FVC is presented for overall participants, and by their peripheral blood eosinophil count (missing, <300 and >=300 cells/uL), smoking history (Lifelong non-smoker, Current and previous smoker) and asthma history (missing, yes, no and unknown).
Time Frame: Baseline (Day 1) and at Month 24
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 529
Liter
  Overall | -0.06 (0.56)
  Peripheral blood EOS: <300 cells/uL: number analyzed (Participants) | 26
  Peripheral blood EOS: <300 cells/uL | 0.02 (0.72)
  Peripheral blood EOS: >=300 cells/uL: number analyzed (Participants) | 17
  Peripheral blood EOS: >=300 cells/uL | -0.13 (0.63)
  Peripheral blood EOS: Missing: number analyzed (Participants) | 486
  Peripheral blood EOS: Missing | -0.06 (0.54)
  Smoking history: Lifelong non-smoker: number analyzed (Participants) | 40
  Smoking history: Lifelong non-smoker | 0.08 (0.55)
  Smoking history: Current smoker: number analyzed (Participants) | 188
  Smoking history: Current smoker | -0.06 (0.59)
  Smoking history: Previous smoker: number analyzed (Participants) | 301
  Smoking history: Previous smoker | -0.08 (0.53)
  Asthma history: No: number analyzed (Participants) | 428
  Asthma history: No | -0.06 (0.56)
  Asthma history: Yes: number analyzed (Participants) | 11
  Asthma history: Yes | 0.07 (0.79)
  Asthma history: Unknown: number analyzed (Participants) | 7
  Asthma history: Unknown | 0.26 (0.52)
  Asthma history: Missing: number analyzed (Participants) | 83
  Asthma history: Missing | -0.11 (0.47)

41. Secondary Outcome: Percentage of Participants With Change in COPD Symptoms at Months 6, 12 and 24 From Baseline
Description: Change in COPD symptoms were evaluated through COPD Assessment Test (CAT) and were categorized as stable symptoms, less symptoms, and more symptoms by comparing with Baseline. Percentage of participants with change in COPD symptoms at Months 6, 12 and 24 from Baseline have been presented. Baseline was considered as Day 1 of inclusion date to the study (Study Day 1). Percentage values are rounded-off.
Time Frame: Baseline (Day 1), Months 6, 12 and 24
Population: as for outcome 13
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 1088
Percentage of participants
  Month 6: Stable symptoms | 77.3
  Month 6: Less symptoms | 15.6
  Month 6: More symptoms | 7.1
  Month 12: Stable symptoms: number analyzed (Participants) | 1016
  Month 12: Stable symptoms | 81.3
  Month 12: Less symptoms: number analyzed (Participants) | 1016
  Month 12: Less symptoms | 10.8
  Month 12: More symptoms: number analyzed (Participants) | 1016
  Month 12: More symptoms | 7.9
  Month 24: Stable symptoms: number analyzed (Participants) | 927
  Month 24: Stable symptoms | 82.6
  Month 24: Less symptoms: number analyzed (Participants) | 927
  Month 24: Less symptoms | 11.0
  Month 24: More symptoms: number analyzed (Participants) | 927
  Month 24: More symptoms | 6.4

42. Secondary Outcome: Change From Baseline in European Quality of Life 5 Dimensions 5 Level (EQ-5D-5L) at Months 12 and 24
Description: EQ-5D-5L is self-assessment questionnaire,consisting of 5 items covering 5 dimensions (mobility,self care,usual activities,pain/discomfort and anxiety/depression). Each dimension is measured by 5-point Likert scale (1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems and 5=extreme problems). Responses for 5 dimensions together formed a 5-figure description of health state (e.g.11111 indicates no problems in all 5 dimensions). Each of these 5 figure health states were converted to a single index score by applying country-specific value set formula that attaches weights to dimensions and levels. Range for EQ-5D-5L index score is -0.594 (worst health) to 1 (full health state). Baseline was considered as Day 1 of inclusion date to the study (Study Day 1). Change from Baseline was calculated as the post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1), Months 12 and 24
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 621
Scores on a scale
  Month 12 | -0.006 (0.222)
  Month 24: number analyzed (Participants) | 528
  Month 24 | 0.003 (0.219)

43. Secondary Outcome: Percentage of Participants Experiencing a Clinically Important Deterioration
Description: Clinically important deterioration was defined as if at least one of the following conditions exists at any point of time during the observational period: decrease (>=100 milliliter [mL]) of FEV1 from Baseline (missing values are treated as no decrease); increase (>2 units) of CAT from Baseline (missing values are treated as no increase); any documented exacerbation; and all-cause mortality. Percentage of participants experiencing a clinically important deterioration during 24 months observation period have been presented. Percentage values are rounded-off.
Time Frame: Up to 24 months
Population: Full Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 1196
Percentage of participants | 53.6

44. Secondary Outcome: Time to First Moderate or Severe Exacerbation
Description: The time to first moderate or severe exacerbation was defined as the duration between onset of first moderate or severe acute exacerbation of COPD from Day 1. Moderate exacerbations are defined as COPD exacerbations that require either systemic corticosteroids and/or antibiotics. Severe exacerbations are defined as those requiring hospitalization (including intubation and admittance to an intensive care unit) or result in death. It was evaluated by Kaplan-Maier analysis.
Time Frame: Up to 24 months
Population: Full Analysis Set.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 1196
Days | NA [NA to NA] — <25% of participants experienced the event within the population. Hence, median and inter-quartiles could not be derived.

45. Secondary Outcome: Time to First Hospitalization
Description: Time to first hospitalization is calculated as the time interval between date of study enrollment (Day 1) and the date of the first hospital admission for a relevant cause. Time to first hospitalization was analyzed using Kaplan-Meier methods.
Time Frame: Up to 24 months
Population: Full Analysis Set.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 1196
Days | NA [NA to NA] — <25% of participants experienced the event within the population. Hence, median and inter-quartiles could not be derived.

46. Secondary Outcome: Time to Death
Description: Time to death is calculated as the duration between date of study enrollment (Day 1) and the date of death of a participant. Time to death was analyzed using Kaplan-Meier methods.
Time Frame: Up to 24 months
Population: Full Analysis Set
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 1196
Days | NA [NA to NA] — <25% of participants experienced the event within the population. Hence, median and inter-quartiles could not be derived.

47. Secondary Outcome: Number of COPD Related Visits
Description: Number of COPD related visits made by participants have been presented and categorized by type of physician (general practitioners and pneumologists).
Time Frame: Up to 24 months
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Number of visits
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 1196
Number of visits
  General practitioners: number analyzed (Participants) | 465
  General practitioners | 5.8 (0.89)
  Pneumologists: number analyzed (Participants) | 731
  Pneumologists | 3.7 (0.89)

48. Secondary Outcome: Mean Annual Rate of Exacerbations Over a 24-month Observation Period Categorized by Physician
Description: The annual rate of exacerbations during the observation period (per participant per year) was assessed. Annualized rate of exacerbations was calculated as Annual exacerbation rate = total number of exacerbation/total person years. Data for mean annual rate of exacerbations categorized by general practitioners and pneumologists have been presented.
Time Frame: Up to 24 months
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Exacerbations per participant per year
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 1196
Exacerbations per participant per year
  General practitioners: number analyzed (Participants) | 465
  General practitioners | 0.182 (0.479)
  Pneumologists: number analyzed (Participants) | 731
  Pneumologists | 0.140 (0.456)

49. Secondary Outcome: Mean Annual Rate of Hospitalization Due to Severe Exacerbation Over a 24-month Observation Period Categorized by Physician
Description: Annualized rate of hospitalization due to severe exacerbations was calculated as Annual hospitalization rate=number of hospitalizations due to severe exacerbations/total person years. Severe exacerbations are defined as COPD exacerbations requiring hospitalization (including intubation and admittance to an intensive care unit) or result in death. Data for mean annual rate of hospitalization due to severe exacerbation categorized by general practitioners and pneumologists have been presented.
Time Frame: Up to 24 months
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Hospitalization per participant per year
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 1196
Hospitalization per participant per year
  General practitioners: number analyzed (Participants) | 465
  General practitioners | 0.027 (0.142)
  Pneumologists: number analyzed (Participants) | 731
  Pneumologists | 0.078 (0.369)

50. Secondary Outcome: Percentage of Participants Categorized by the Site Localization of Physician and by Type of Physician
Description: Percentage of participants have been categorized according to the site localization (East, North, South, and West Germany) of physician and type of physician (general practitioners and pneumologists). Percentage values are rounded-off.
Time Frame: Up to 24 months
Population: as for outcome 13
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 1196
Percentage of participants
  General practitioners: East Germany: number analyzed (Participants) | 465
  General practitioners: East Germany | 9.2
  General practitioners: North Germany: number analyzed (Participants) | 465
  General practitioners: North Germany | 29.2
  General practitioners: South Germany: number analyzed (Participants) | 465
  General practitioners: South Germany | 29.5
  General practitioners: West Germany: number analyzed (Participants) | 465
  General practitioners: West Germany | 32.0
  Pneumologists: East Germany: number analyzed (Participants) | 731
  Pneumologists: East Germany | 33.0
  Pneumologists: North Germany: number analyzed (Participants) | 731
  Pneumologists: North Germany | 7.8
  Pneumologists: South Germany: number analyzed (Participants) | 731
  Pneumologists: South Germany | 7.5
  Pneumologists: West Germany: number analyzed (Participants) | 731
  Pneumologists: West Germany | 51.7

51. Secondary Outcome: Mean Annual Rate of Exacerbations Over a 24-month Observation Period Categorized by Type of Physician and by Peripheral Blood Eosinophil Count, Smoking Status and Asthma History
Description: The annual rate of exacerbations during the observation period (per participant per year) was assessed. Annualized rate of exacerbations was calculated as Annual exacerbation rate = total number of exacerbation/total person years. Data for mean annual rate of exacerbations is presented by smoking status (Lifelong non-smoker, Current and previous smoker), peripheral blood eosinophil count (missing, <300 and >=300 cells/uL), and asthma history (missing, yes, no and unknown). Data was also categorized by the type of physician (general practitioners and pneumologists).
Time Frame: Up to 24 months
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Exacerbations per participant per year
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 1196
Exacerbations per participant per year
  General practitioners: Smoking status- Lifelong non-smoker: number analyzed (Participants) | 53
  General practitioners: Smoking status- Lifelong non-smoker | 0.158 (0.559)
  General practitioners: Smoking status- Current smoker: number analyzed (Participants) | 160
  General practitioners: Smoking status- Current smoker | 0.143 (0.336)
  General practitioners: Smoking status- Previous smoker: number analyzed (Participants) | 252
  General practitioners: Smoking status- Previous smoker | 0.211 (0.535)
  General practitioners: Eosinophil count- Missing: number analyzed (Participants) | 433
  General practitioners: Eosinophil count- Missing | 0.187 (0.493)
  General practitioners: Eosinophil count- <300 cells/uL: number analyzed (Participants) | 24
  General practitioners: Eosinophil count- <300 cells/uL | 0.072 (0.189)
  General practitioners: Eosinophil count- >=300 cells/uL: number analyzed (Participants) | 8
  General practitioners: Eosinophil count- >=300 cells/uL | 0.119 (0.216)
  General practitioners: Asthma history- Missing: number analyzed (Participants) | 9
  General practitioners: Asthma history- Missing | 0.252 (0.637)
  General practitioners: Asthma history- No: number analyzed (Participants) | 387
  General practitioners: Asthma history- No | 0.159 (0.433)
  General practitioners: Asthma history- Yes: number analyzed (Participants) | 58
  General practitioners: Asthma history- Yes | 0.439 (0.732)
  General practitioners: Asthma history- Unknown: number analyzed (Participants) | 11
  General practitioners: Asthma history- Unknown | 0.386 (0.711)
  Pneumologists: Smoking status- Lifelong non-smoker: number analyzed (Participants) | 53
  Pneumologists: Smoking status- Lifelong non-smoker | 0.099 (0.331)
  Pneumologists: Smoking status- Current smoker: number analyzed (Participants) | 294
  Pneumologists: Smoking status- Current smoker | 0.080 (0.270)
  Pneumologists: Smoking status- Previous smoker: number analyzed (Participants) | 384
  Pneumologists: Smoking status- Previous smoker | 0.191 (0.565)
  Pneumologists: Eosinophil count- Missing: number analyzed (Participants) | 669
  Pneumologists: Eosinophil count- Missing | 0.118 (0.387)
  Pneumologists: Eosinophil count- <300 cells/uL: number analyzed (Participants) | 41
  Pneumologists: Eosinophil count- <300 cells/uL | 0.619 (1.077)
  Pneumologists: Eosinophil count- >=300 cells/uL: number analyzed (Participants) | 21
  Pneumologists: Eosinophil count- >=300 cells/uL | 0.302 (0.812)
  Pneumologists: Asthma history- Missing: number analyzed (Participants) | 5
  Pneumologists: Asthma history- Missing | 0.137 (0.454)
  Pneumologists: Asthma history- No: number analyzed (Participants) | 536
  Pneumologists: Asthma history- No | 0.146 (0.456)
  Pneumologists: Asthma history- Yes: number analyzed (Participants) | 135
  Pneumologists: Asthma history- Yes | 0.048 (0.156)
  Pneumologists: Asthma history- Unknown: number analyzed (Participants) | 55
  Pneumologists: Asthma history- Unknown | 0.116 (0.532)

52. Secondary Outcome: Number of Participants Who Had Pneumonia and Cardiovascular Events
Description: Number of participants who had pneumonia and cardiovascular events have been presented.
Time Frame: Up to 24 months
Population: Safety Analysis Set included all participants who signed the ICF, met all inclusion criteria and none of the exclusion criteria, and completed visit 1. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the Overall Number of Participants Analyzed field.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 1196
Participants
  Pneumonia events | 22
  Cardiovascular events | 23

53. Secondary Outcome: Number Needed to Treat for Benefit (NNTB) for SITT Participants Compared to Non SITT With Respect to Exacerbations, Pneumonia, and Cardiovascular Events
Description: NNTB is a metric used to assess the benefit of treatment. It indicates how many participants need to be treated to achieve one additional beneficial outcome with respect to exacerbations, pneumonia, and cardiovascular events. NNTB is presented as number of participants and is presented at Days 90 and 365 for participants on SIIT compared to non SITT. A participant is classified as SITT, if the treatment is SITT continuously for the first 365 days of observation.
Time Frame: Days 90 and 365
Population: Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 1196
Participants
  Day 90: NNTB with respect to Exacerbations | 58
  Day 365: NNTB with respect to Exacerbations | 15
  Day 90: NNTB with respect to Pneumonia | NA — Data could not be derived because there was a harm and no benefit of treatment.
  Day 365: NNTB with respect to Pneumonia | NA — Data could not be derived because there was a harm and no benefit of treatment.
  Day 90: NNTB with respect to Cardiovascular events | 1042
  Day 365: NNTB with respect to Cardiovascular events | NA — Data could not be derived because there was a harm and no benefit of treatment.

54. Secondary Outcome: Number Needed to Treat for Benefit (NNTB) for MITT Participants Compared to Non MITT With Respect to Exacerbations, Pneumonia, and Cardiovascular Events
Description: NNTB is a metric used to assess the benefit of treatment. It indicates how many participants need to be treated to achieve one additional beneficial outcome with respect to exacerbations, pneumonia, and cardiovascular events. NNTB is presented as number of participants and is presented at Days 90 and 365 for participants on MITT compared to non MITT. A participant is classified as MITT, if the treatment is MITT continuously for the first 365 days of observation.
Time Frame: Days 90 and 365
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 1196
Participants
  Day 90: NNTB with respect to Exacerbations | 131
  Day 365: NNTB with respect to Exacerbations | 25
  Day 90: NNTB with respect to Pneumonia | 146
  Day 365: NNTB with respect to Pneumonia | 91
  Day 90: NNTB with respect to Cardiovascular events | 203
  Day 365: NNTB with respect to Cardiovascular events | 98

55. Secondary Outcome: Number Needed to Treat for Benefit (NNTB) With Respect to Exacerbations, Pneumonia, and Cardiovascular Events for Participants Whose Triple Therapies Interrupted by ICS and/or LAMA "Off/on" Periods Compared to Other Triple Therapies
Description: NNTB is a metric used to assess the benefit of treatment. It indicates how many participants need to be treated to achieve one additional beneficial outcome with respect to exacerbations, pneumonia, and cardiovascular events. NNTB is presented as number of participants and is presented at Days 90 and 365 for participants whose triple therapies were interrupted by ICS and/or LAMA "off/on" periods compared to other triple therapies.
Time Frame: Days 90 and 365
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 1196
Participants
  Day 90: NNTB with respect to Exacerbations | NA — Data could not be derived because there was a harm and no benefit of treatment.
  Day 365: NNTB with respect to Exacerbations | NA — Data could not be derived because there was a harm and no benefit of treatment.
  Day 90: NNTB with respect to Pneumonia | 163
  Day 365: NNTB with respect to Pneumonia | 41
  Day 90: NNTB with respect to Cardiovascular events | 226
  Day 365: NNTB with respect to Cardiovascular events | 61

56. Secondary Outcome: Number Needed to Treat for Benefit (NNTB) With Respect to Exacerbations, Pneumonia, and Cardiovascular Events for Participants With Switch of Triple Therapies Between SITT and MITT Compared to no Switch
Description: NNTB is a metric used to assess the benefit of treatment. It indicates how many participants need to be treated to achieve one additional beneficial outcome with respect to exacerbations, pneumonia, and cardiovascular events. NNTB is presented as number of participants and is presented at Days 90 and 365 for participants whose triple therapies were switched between SITT and MITT compared to no switch. A participants is classified as switch, if there is no de-escalation of therapy, but at least one switch between SITT and MITT within the first 365 days of observation.
Time Frame: Days 90 and 365
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
Number analyzed (Participants) | 1196
Participants
  Day 90: NNTB with respect to Exacerbations | NA — Data could not be derived because there was a harm and no benefit of treatment.
  Day 365: NNTB with respect to Exacerbations | NA — Data could not be derived because there was a harm and no benefit of treatment.
  Day 90: NNTB with respect to Pneumonia | 159
  Day 365: NNTB with respect to Pneumonia | 40
  Day 90: NNTB with respect to Cardiovascular events | NA — Data could not be derived because there was a harm and no benefit of treatment.
  Day 365: NNTB with respect to Cardiovascular events | NA — Data could not be derived because there was a harm and no benefit of treatment.

ADVERSE EVENTS:
Time Frame: All-cause mortality, non-serious drug-related adverse events and serious adverse events (SAEs) were collected up to 24 months
Description: Only all-cause mortality, SAEs and non-serious drug-related adverse events were collected, but not all non-SAEs. Safety analysis set included all participants who signed the ICF, met all inclusion criteria and none of the exclusion criteria, and completed visit 1. 16 participants from enrolled population were with incomplete documentation, hence were not included in Safety analysis set.
Arm/Group | Participants With Chronic Obstructive Pulmonary Disease (COPD)
All-Cause Mortality (participants affected / at risk) | 51/1196
Serious Adverse Events (participants affected / at risk) | 142/1196
Other Adverse Events (participants affected / at risk) | 16/1196
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Chronic Obstructive Pulmonary Disease (COPD) (N=1196)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 18
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 2
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1
Tracheomalacia (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Infections and infestations) | 19
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 3
COVID-19 (Infections and infestations) | 2
Diverticulitis (Infections and infestations) | 2
Influenza (Infections and infestations) | 2
Atypical mycobacterial infection (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Pneumonia aspiration (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Tick-borne viral encephalitis (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Death (General disorders) | 20
Multiple organ dysfunction syndrome (General disorders) | 2
Chest pain (General disorders) | 1
Gait disturbance (General disorders) | 1
Impaired healing (General disorders) | 1
Cardiac failure (Cardiac disorders) | 10
Atrial fibrillation (Cardiac disorders) | 6
Acute myocardial infarction (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Cardiac disorder (Cardiac disorders) | 1
Cardiac failure chronic (Cardiac disorders) | 1
Cor pulmonale chronic (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Elastofibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oropharyngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancoast's tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Fall (Injury, poisoning and procedural complications) | 5
Humerus fracture (Injury, poisoning and procedural complications) | 2
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2
Alcohol poisoning (Injury, poisoning and procedural complications) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Skin laceration (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Cerebrovascular accident (Nervous system disorders) | 5
Transient ischaemic attack (Nervous system disorders) | 2
Aphasia (Nervous system disorders) | 1
Cerebral ischaemia (Nervous system disorders) | 1
Dementia Alzheimer's type (Nervous system disorders) | 1
Senile dementia (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Abdominal hernia (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Duodenal perforation (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal vascular malformation haemorrhagic (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1
Muscle swelling (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 2
Aortic aneurysm (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Marasmus (Metabolism and nutrition disorders) | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 1
Panic attack (Psychiatric disorders) | 1
Psychotic disorder (Psychiatric disorders) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Normocytic anaemia (Blood and lymphatic system disorders) | 1
Vertigo positional (Ear and labyrinth disorders) | 1
Diplopia (Eye disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Chronic Obstructive Pulmonary Disease (COPD) (N=1196)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Eczema (Skin and subcutaneous tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Glossodynia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Oral candidiasis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Palpitations (Cardiac disorders) | 1
Oedema peripheral (General disorders) | 1
C-reactive protein abnormal (Investigations) | 1
International normalised ratio abnormal (Investigations) | 1
Weight decreased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-02-16): https://cdn.clinicaltrials.gov/large-docs/11/NCT04657211/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-25): https://cdn.clinicaltrials.gov/large-docs/11/NCT04657211/SAP_001.pdf